CLINICAL TRIAL: NCT00908700
Title: Phase III Pilot Study - Left Atrial Appendage Occlusion Study
Brief Title: Left Atrial Appendage Occlusion Study II
Acronym: LAAOSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: McMaster University (Other); Sunnybrook Health Sciences Centre (Other); London Health Sciences Centre (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Richard Whitlock, Cardiovascular Surgeon, Department of Surgery, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAAOSII
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial fibrillation; Stroke; left atrial appendage; Re-exploration for bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occlusion arm (Experimental): Surgical intervention: Occlusion of the left atrial appendage (LAA) using 'cut-and-sew' technique appendage occlusion.
  Interventions: Procedure: Surgical occlusion of the left atrial appendage
- Medical arm (Active Comparator): Medical arm: The comparator is best medical practice for atrial fibrillation related stroke prevention as per guidelines.
  Interventions: Procedure: Best medical practice

INTERVENTIONS:
Procedure: Surgical occlusion of the left atrial appendage — Study intervention: Within the trial, occlusion must be performed using either amputation and closure (cut and sew) or stapler device.
  Arms: Occlusion arm
Procedure: Best medical practice — Best medical practice for atrial fibrillation related stroke prevention as per guidelines.
  Arms: Medical arm

SUMMARY:
A pilot, multicentre randomized controlled study of surgical left atrial occlusion (LAA) in 50 patients with atrial fibrillation/flutter undergoing cardiac surgery requiring cardiopulmonary bypass with additional risk factors for late stroke.

Patients will be enrolled and randomized to undergo LAA exclusion and aspirin therapy or best medical therapy as per guidelines.

Main research questions:

1. Can successful occlusion of the LAA be safely achieved by cut and sew or stapler techniques?
2. In patients with atrial fibrillation with 2 or more risk factors for stroke, will removal of the left atrial appendage (LAA) and aspirin therapy reduce the risk of systemic embolic events and major bleeding compared to warfarin?

DETAILED DESCRIPTION:
The number one cause of disability and the 3rd leading cause of death in patients with atrial fibrillation (AF) is stroke. Echocardiographic studies suggest that the predominant source of stroke in AF is the left atrial appendage (LAA). At present, there are no sufficiently powered trials to answer whether removal of the LAA can reduce the risk of systemic embolic events.

LAAOS pilot study will recruit 50 participants undergoing open-heart surgery in 5 Canadian academic cardiac surgery centers. The study will inform the feasibility of conducting a large RCT and will provide information of the efficacy and safety of appendage occlusion technique. From this study we envision a a large international randomized controlled trial (LAAOS II) to determine the impact of left atrial appendage occlusion on the composite outcome of stroke and non-central nervous system systemic embolic events in at risk patients with atrial fibrillation undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing any cardiac surgical procedure with the use of cardiopulmonary bypass
* A history of ECG-documented atrial fibrillation with prior stroke or TIA, or at least two of the following risk factors:

  * age => 65 years
  * hypertension
  * diabetes mellitus, or
  * heart failure/left ventricular ejection fraction < 50%

Exclusion Criteria:

* Patients in whom surgical AF ablation (MAZE or otherwise) is planned
* Planned "off-pump" surgery
* Planned implantation of a mechanical valve
* Heart transplant, complex congenital heart surgery, and ventricular assist device insertion, reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Demonstration of efficacy of cut-and-sew and stapler technique of appendage occlusion by intraoperative transesophageal echocardiography, central adjudication. | Outcomes will be measured at discharge, 4-8 weeks post-op and long term (1 to 4 years)

SECONDARY OUTCOMES:
Demonstration of study feasibility, procedure safety, including rate of post-operative re-exploration for bleeding. | Outcomes will be measured at discharge, 4-8 weeks post-op and long term (1 to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada